CLINICAL TRIAL: NCT02902848
Title: Evaluation of the Validity of the Prothrombin Time Internation Normalised Ratio (PT/INR) Measured at the point-of Care on the Arterial Bloodline of Haemodialysis Extracorporeal Blood Flow
Acronym: COAGHEMO
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: COAGHEMO
Record Dates: First submitted 2016-09-08; First posted 2016-09-16 (Estimated); Last update posted 2016-09-16 (Estimated); Status verified 2016-09

CONDITIONS: Haemodialysis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
The purpose of this study is to evaluate the INR value of hemodialyzed patient coagulation state (prothrombin time) measured inside the therapeutical zone and thanks to a portable monitor. The values obtained at the point of care will be compared to the standard biological assessment.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18
* Haemodialyzed patient whose INR needs to be monitored
* Patient not objecting to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The population of the study is the patients under haemodialysis treatment, who need INR monitoring
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2015-03; Primary Completion 2017-03 (Estimated)

PRIMARY OUTCOMES:
correlation ratio between point-of-care PT/INR value and standard laboratory assessement | 5 months

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Brest, Brest, France